CLINICAL TRIAL: NCT06275074
Title: Effects of Dry Needling and Therapeutic Exercise on Sleep in Individuals With Chronic Neck Pain and Sleep Disturbance - A Pilot Study
Brief Title: Dry Needling and Therapeutic Exercise on Sleep in Individuals With Chronic Neck Pain and Sleep Disturbance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ray M. Lunasin, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 23-007716
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Neck Pain; Sleep Disturbance
Keywords: Needling; Sleep Disturbance; Chronic pain; Neck Pain; Actigraphy; Physical Therapy; Feasibility
MeSH Terms: conditions — Neck Pain; Parasomnias; Chronic Pain | interventions — Dry Needling; Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group assignment of participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling and Therapeutic Exercise (Experimental)
  Interventions: Procedure: Dry Needling; Other: Therapeutic Exercise
- Therapeutic Exercise Alone (Active Comparator)
  Interventions: Other: Therapeutic Exercise

INTERVENTIONS:
Procedure: Dry Needling — Insertion of filiform needles into cervicothoracic multifidi, upper trapezius, and suboccipital muscles
  Arms: Dry Needling and Therapeutic Exercise
Other: Therapeutic Exercise — Therapeutic exercise program provided to all participants with the aim of addressing periscapular strength and postural edurance.

SUMMARY:
Feasibility study investigating the effects of dry needling on individuals with chronic neck pain and sleep disturbance.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine the feasibility of a large randomized clinical trial (RCT) which aims to investigate the effects of dry needling (DN) in addition to therapeutic exercise (TE) on sleep duration and quality in patients with chronic neck pain (CNP) and sleep disturbance (SD). Specifically, the objective is to explore feasibility of a study protocol and examine the preliminary data of a small sample size for the effectiveness of DN and TE for individuals with CNP and SD to determine effect size of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain lasting greater than 3 months 28,29
* Age: 18-75 years
* Presence of sleep disturbance - to be defined as a score ≥ 8 on the Insomnia Severity Index
* Ability to understand study procedures and to comply with them for the entire length of the study

Exclusion Criteria:

* Previous surgery to the neck or thoracic spine
* Central nervous system disorders
* Systemic joint disease (e.g. rheumatoid arthritis)
* Infection
* Cancer
* Raynaud's disease
* Pregnancy
* Immunocompromised disease (e.g., diabetes mellitus, HIV, AIDS, lupus)
* Insufficient English-language skills to complete all questionnaires.
* Contraindications to dry needling:

  * Presence of needle phobia
  * History of abnormal reaction to needling or injection
  * History of bleeding disorder (e.g., current anticoagulant therapy or known thrombocytopenia)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Participant retention rate | 1 year
  One variable to be assessed to determine feasibility is retention rate of participants recruited and enrolled. The retention rate of participants will be calculated as follows: Retention rate = (Number of patients completing the study / Number of patients initially enrolled) x 100. Feasibility will be determined with 4-week attrition rate is less than 20%
Participant intervention adherence | 1 year
  One variable to be assessed to determine feasibility is intervention adherence. Adherence to therapeutic exercise program given to all participants will be assessed with an exercise diary to be completed by the participants to track exercise compliance. A new diary will be provided on a weekly basis to maintenance of records.
Number of adverse responses to treatment | 1 year
  Occurrence of adverse responses to treatment will be accounted for at each subsequent visit after initial treatment administered (visits 3-6). Patients will be asked to complete an intake form that will inquire about their experience post-intervention and provide examples of common adverse responses to determine if such events occurred for each respective participant.

SECONDARY OUTCOMES:
Sleep Duration | 5 weeks
  Total sleep time and Sleep latency via wrist actigraphy
Sleep Quality | 13 weeks
  Sleep quality will be measured with the use of the Pittsburgh Sleep Quality Index (PSQI). There are seven components that range in scores of 0-3. Total scores range from 0-21 with higher scores indicating worse sleep quality.

OTHER OUTCOMES:
Disability Level | 13 weeks
  Disability level will be measured with the Neck Pain Disability Index (NDI). There are ten questions with a range of scores of 0-5. Total possible scores range from 0-50 or 0%-100% with higher scores indicating greater disability level.
Pain Level | 13 weeks
  Pain level will be measured using the numerical pain rating scale (NPRS). It is an 11-point numeric scale ranging from '0' representing "no pain" to '10' representing "worst pain imaginable."

CONTACTS AND LOCATIONS:
Overall Officials: Ray Lunasin, P.T., D.P.T., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic - Motion Analysis Lab, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trial webpage of study — https://www.mayo.edu/research/clinical-trials/cls-20563436